CLINICAL TRIAL: NCT07215624
Title: Surgical Thromboprophylaxis Practices in Oncology Patients Within the NCORP Network (STOP-VTE)
Brief Title: Surgical Thromboprophylaxis Practices in Oncology Patients Within the NCORP Network, STOP-VTE Study
Acronym: STOP-VTE
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00138219; NCI-2025-06376 (Other: NCI Trial Identifier); WF-2502CD (Other: Lead Organization Identifier); WF-2502CD (Other: DCP Identifier); WF-2502CD (Other: CTEP Identifier)
Record Dates: First submitted 2025-09-29; First posted 2025-10-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Malignant Digestive System Neoplasm; Malignant Female Reproductive System Neoplasm; Malignant Genitourinary System Neoplasm
MeSH Terms: conditions — Gastrointestinal Neoplasms; Urogenital Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Observational Part 1: Surgeons and APPs complete a survey on study. After completion of surgeon or APP survey, site contact person or CCDR lead complete site surveys on study.
  Interventions: Other: Non-Interventional Study
- Observational Part 2: Subset of surgeons and APPs from Part 1 complete a semi-structured interview on study.
  Interventions: Other: Non-Interventional Study
- Observational Part 3: Site contact person or CCDR lead complete a survey to identify a EHR Report Specialist on study. EHR Report Specialist performs an EHR Data Extraction and provides feedback on the process in a survey.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study
  Groups: Observational Part 1
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study
  Groups: Observational Part 2
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study
  Groups: Observational Part 3

SUMMARY:
This study evaluates the use of extended venous thromboembolism prophylaxis (ePPx) following abdominopelvic cancer surgery within the NCI Community Oncology Research Program (NCORP) network, targeting surgeons and surgical advanced practice providers (APPs).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate self-reported utilization of guideline concordant extended venous thromboembolism (VTE) prophylaxis (ePPx) following abdominopelvic cancer surgery within a sample of surgeons practicing within NCORP based on the Part 1 surgeon survey.

SECONDARY OBJECTIVES:

I. Evaluate site factors (e.g., proportion of publicly insured patients, proportion of Black patients, presence of a medical school, NCI designation) and surgeon factors (e.g., fellowship training, years in practice) associated with surgeon self-reported guideline concordant ePPx utilization (Part 1).

II. Conduct semi-structured interviews among a subset of surgeons and surgical APPs to assess: 1) Barriers/facilitators toward ePPx after cancer surgery and 2) Acceptability of clinical decision support tools to support VTE prophylaxis prescribing (Part 2).

III. Extract EHR data from select practices to assess the feasibility of query-based electronic health record (EHR) data extraction for identification of (i) patients undergoing cancer surgery, and (ii) prescription of guideline concordant ePPx among eligible patients (Part 3).

OUTLINE: This is an observational study.

PART 1: Surgeons and APPs complete a survey on study. After completion of surgeon or APP survey, site contact person or Cancer Care Delivery Research (CCDR) lead complete site surveys on study.

PART 2: A subset of surgeons and APPs from part 1 complete a semi-structured interview on study.

PART 3: Site contact person or CCDR lead complete a survey to identify a EHR Report Specialist on study. EHR Report Specialist performs an EHR Data Extraction and provides feedback on the process in a survey.

ELIGIBILITY:
Inclusion Criteria:

SURGEON ELIGIBILITY CRITERIA FOR OPEN STEP 0 ENROLLMENT:

* Any surgeon performing gastrointestinal, genitourinary, or gynecologic cancer surgery within an NCORP site, including general surgeons, surgical specialists, urologists, and gynecologists. Surgeons do not need to be involved in research or have a Cancer Therapy Evaluation Program Identification (CTEP ID) to participate in this study

SURGICAL APP ELIGIBILITY CRITERIA FOR OPEN STEP 0 ENROLLMENT:

* APPs providing postoperative care to patients operated by surgeons performing gastrointestinal, genitourinary, or gynecologic cancer surgery within an NCORP site, including general surgeons, surgical specialists, urologists, and gynecologists. Surgical APPs do not need to be involved in research or have a CTEP ID to participate in this study

SURGEON ELIGIBILITY CRITERIA FOR OPEN STEP 1 ENROLLMENT:

* Must have completed the STOP-VTE Survey - Surgeon electronically (preferred) or on paper and have it transferred to Research Electronic Data Capture (REDCap) by the contact person(s)

SURGICAL APP ELIGIBILITY CRITERIA FOR OPEN STEP 1 ENROLLMENT:

* Must have completed the STOP-VTE Survey - APP electronically (preferred) or on paper and have it transferred to REDCap by the contact person(s)

SITE ELIGIBILITY PART 1-SITE ENROLLMENT IN OPEN:

* Have at least one eligible surgeon or surgical APP who completed the STOP-VTE Survey - Surgeon/APP

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This multi-part study employs a mixed-methods design to evaluate the utilization of ePPx following abdominopelvic cancer surgery within the NCORP network. Part 1 involves a cross-sectional survey of at least 100 surgeons/APPs from at least 25 NCORP sites to evaluate practice patterns related to ePPx. Part 2 utilizes purposive sampling to conduct interviews with 11-25 surgeons/APPs from Part 1 to obtain granular detail about barriers and facilitators to guideline concordant utilization of ePPx. Part 3 will purposively sample 6 practices identified in Part 1 to evaluate the feasibility of EHR queries to assess ePPx utilization.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported utilization of guideline concordant ePPx for surgeons (Part 1) | After 1 year from start of Part 1
  Will apply only to surgeons completing the Part 1 survey. Will be defined as answering "Yes, all cases or almost all cases" on the survey question asking about prescription of ePPx after discharge. The proportion of surgeons self-reporting utilization of guideline concordant ePPx will be estimated and reported along with an exact 95% confidence interval.

SECONDARY OUTCOMES:
Self-reported utilization of guideline concordant ePPx for surgeons within strata defined by site and surgeon factors (Part 1) | After 1 year from start of Part 1
  Self reported utilization as defined above for the primary outcome measure will be reported within strata defined by:
  * Site factors (e.g., proportion of publicly insured patients, proportion of Black patients, presence of a medical school, NCI designation)
  * Surgeon factors (e.g., fellowship training, years in practice)
Barriers and facilitators toward ePPx after cancer surgery, and acceptability of clinical decision support tools to support VTE prophylaxis prescribing (Part 2) | After 6 months from start of Part 2
  Themes from qualitative interviews by surgeons and APPs
Feasibility (i.e., proportion of practices able to provide data) of EHR queries from selected practices to inform future trial (Part 3) | After 6 months from start of Part 3
  Considered feasible if at least 4 of the 6 practices who agreed to participate are able to provide data on both patients undergoing cancer surgery and prescription of guideline concordant ePPx among eligible patients

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Lesser, MD, Study Chair — Wake Forest University Health Sciences
Locations (28):
- United States (28):
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Blank Children's Hospital, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Wake Forest NCORP Research Base, Winston-Salem, North Carolina
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Charleston Oncology North Charleston, Charleston, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest NCORP Research Base is committed to following the NIH Statement on Sharing Research Data (http://grants.nih.gov/grants/guide/notice-files/NOT-OD-03-032.html). As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI NCTN/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials to https://nctn-data-archive.nci.nih.gov/. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide. De-identified data from studies not covered by the agreement (e.g., phase II and observational studies) will be made available upon request. All data files will be de-identified. De-identification procedures will meet the HIPAA criteria as detailed in the Code of Federal Regulations, Part 45, Section 164.514.
Time Frame: 6 months after publication for a 2 year duration
Access Criteria: upon request to NCORP@wakehealth.edu